CLINICAL TRIAL: NCT07157475
Title: Ocena powikłań Naczyniowych u pacjentów Poddanych Rewaskularyzacji Obwodowej: wpływ inhibitorów SGLT-2 The Assessment of Vascular Complications in Patients Undergoing Peripheral Revascularization: The Impact of SGLT-2 Inhibitors
Brief Title: Vascular Complications in Patients Undergoing Peripheral Revascularization and Taking SGLT-2 Inhibitors
Status: Recruiting | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Collaborators: Poznan University of Medical Sciences (Other); Military Institute of Medicine National Research Institute (Unknown)
Responsible Party: Principal Investigator, Edyta Sutkowska, M.D., Ph.D., Wroclaw Medical University
Other Study IDs: BW-24/2025
Record Dates: First submitted 2025-08-18; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Arterial Disease(PAD)
Keywords: flozins; SGLT2i; peripheral arterial disease; revascularisation; MACE; MALE
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Therapeutics; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients after vascular surgery treated with flozins: Patients aged ≥18 years who have undergone vascular surgery (either open or minimally invasive procedures) and, for any reason, were treated with SGLT2 inhibitors ("flozins") during the one-year follow-up period after the procedure.
  Interventions: Drug: Treatment with SGLT2 inhibitors (flozins)
- Patients after vascular surgery with no exposure to flozins (controls): Patients aged ≥18 years who have undergone vascular surgery (either open or minimally invasive procedures) and were not exposed to SGLT2 inhibitors ("flozins") during the one-year follow-up period after the procedure.

INTERVENTIONS:
Drug: Treatment with SGLT2 inhibitors (flozins) — Patients received SGLT2 inhibitors (empagliflozin, dapagliflozin, canagliflozin) as part of their routine clinical care during the 12-month follow-up period after elective or urgent lower limb revascularization procedures. The study does not assign treatment; medication use occurred independently of the study protocol.
  Groups: Patients after vascular surgery treated with flozins

SUMMARY:
The study is observational and involves patients (pts) with peripheral arterial occlusive disease (PAD) who have undergone lower limb revascularization procedures. Patients who are at least one year post-procedure will be contacted by phone and asked whether any cardiovascular complications occurred during that period, specifically major adverse cardiovascular events (MACE) or major adverse limb events (MALE), and whether they had been taking sodium-glucose co-transporter 2 inhibitors (SGLT2-i, "flozins") during the year following the procedure. The results from the group of pts who, for any reason, received SGLT2-i treatment after the vascular procedure (including those who had initiated treatment before surgery) will be compared to the results from the group of patients who did not receive such treatment, with regard to the occurrence of the aforementioned complications.

DETAILED DESCRIPTION:
Project Objective: To assess the impact of SGLT2 inhibitors (SGLT2-i) on vascular complications in patients undergoing peripheral revascularization.

Specific Objective: To evaluate the incidence of 3-point MACE* (Major Adverse Cardiac Events) and MALE** (Major Adverse Limb Events) following vascular surgical procedures (both open and minimally invasive), performed in patients treated with SGLT2- i vs controls ( non-treated pts).

Observation Period: One year - assessment at 30 days, 3 months, and 1 year post-procedure.

Definitions for:

* MACE = Non-fatal myocardial infarction (MI),Non-fatal stroke involving the central nervous system (CNS), Cardiovascular death

** MALE = Untreated restenosis or deterioration in patency of a previously revascularized vessel , Reintervention in the revascularized segment due to impaired patency, Amputation (either above or below the knee) of the revascularized limb.

Demographic and clinical data will be obtained from the medical records of patients hospitalized in three vascular surgery departments (Wrocław, Poznań, Warsaw), while information regarding MACE , MALE, and the use of SGLT2-i will be collected via telephone interviews with the patients (or their family members, if the patient is deceased).

The number of MACE and MALE incidents during the year following the procedure will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral vascular procedure ( Conventional surgical procedure or minimally invasive procedure) due to acute or chronic ischemia
* Use of SGLT2 inhibitors (applies only to the group exposed to flozins) for at least 3 months prior to the vascular procedure (the indication for initiating the drug is irrelevant: chronic kidney disease [CKD] / cardiac reasons / diabetes), or immediately after the vascular procedure
* Ability to determine the patient's outcomes within a minimum of 30 days up to 1 year following the vascular procedure

Exclusion Criteria:

* Vascular injury as the reason for the procedure
* Amputation due to causes other than ischemia (e.g., cancer, neuropathy, trauma without coexisting ischemia)
* Planned revascularization procedure other than for the lower limbs at the time of hospital discharge (e.g., coronary or carotid arteries)
* Planned ischemia-related amputation or reoperation of the operated limb at the time of hospital discharge
* Planned other major surgical procedure with high cardiovascular risk at the time of hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The analyzed cases will involve patients from three major vascular clinics located in Wrocław, Poznań, and Warsaw.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE (Major Adverse Cardiovascular Events) and MALE (Major Adverse Limb Events)-Number of Participants Experiencing MACEor MALE | 12 months from the vascular intervention
  MACE is defined as a composite of : Non-fatal myocardial infarction (MI); Non-fatal stroke involving the central nervous system (CNS); or Cardiovascular death MALE is defined as a composite of : Untreated loss or deterioration of patency in a previously revascularized vessel; Repeat intervention in a revascularized segment due to impaired patency, or Amputation (above or below the knee) of the revascularized limb Unit of Measure: Number of participants with at least one event

SECONDARY OUTCOMES:
Non-fatal Myocardial Infarction (MI) | 12 months from the vascular intervention
  Non-fatal myocardial infarction (MI), Unit of Measure: Number of participants
  Non-fatal stroke involving the central nervous system (CNS)
  Cardiovascular death
  Untreated loss or deterioration of patency in a previously revascularized vessel
  Repeat intervention in a revascularized segment due to impaired patency
  Amputation (above or below the knee) of the revascularized limb
Non-fatal Stroke Involving the Central Nervous System (CNS) | 12 months from the vascular intervention
  Non-fatal Stroke Involving the Central Nervous System (CNS), Unit of Measure: Number of participants
Cardiovascular Death | 12 months from the vascular intervention
  Cardiovascular Death, Unit of Measure: Number of participants
Loss or Deterioration of Patency in a Previously Revascularized Vessel | 12 months from the vascular intervention
  Loss or Deterioration of Patency in a Previously Revascularized Vessel, Unit of Measure: Number of participants
Repeat intervention in a revascularized segment due to impaired patency | 12 months from the vascular intervention
  Repeat intervention in a revascularized segment due to impaired patency; Unit of Measure: Number of participants and number of limbs
Amputation of the revascularized limb | 12 months from the vascular intervention
  Amputation (above or below the knee) of the revascularized limb; Unit of Measure: Number of participants and number of limbs

OTHER OUTCOMES:
Additional secondary endpoint- Surgical site infection (SSI) | 12 months from vascular intervention
  Surgical site infection occurring after the index vascular intervention. Unit of Measure: Number of participants
Additional secondary endpoint- Significant bleeding | 12 months from vascular intervention
  Clinically significant bleeding events as assessed by treating physician (according to established clinical criteria). Unit of Measure: Number of participants
Additional secondary endpoint- Kidney injury | 12 months from vascular intervention
  Acute kidney injury occurring after vascular intervention, defined according to KDIGO (Kidney Disease: Improving Global Outcomes) criteria. Unit of Measure: Number of participants
Additional secondary endpoint- Reintervention in the Same Vascular Segment | 12 months from vascular intervention
  Readmission and repeat procedure in the same vascular segment due to impaired patency. Unit of Measure: Number of participants and number of limbs
Additional secondary endpoint- Foot Necrosis | 12 months from vascular intervention
  Development of necrosis in the treated limb within the study period. Unit of Measure: Number of participants and number of limbs
Additional secondary endpoint- Minor Amputation | 12 months from vascular intervention
  Minor amputation defined as amputation within the foot (below the ankle). Unit of Measure: Number of participants and number of limbs
Additional secondary endpoint- Heart Failure Hospitalization | 12 months from vascular intervention
  Hospital admission with a primary diagnosis of heart failure. Unit of Measure: Number of participants

CONTACTS AND LOCATIONS:
Overall Officials: Edyta Sutkowska, Ph.D, Study Chair — Wroclaw Medical University
Locations (1):
- Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol
Time Frame: Individual participant data (de-identified) and supporting documents will be available upon reasonable request from qualified researchers, starting 6 months after publication of the primary results and for a period of 5 years.
Access Criteria: Anonymized individual participant data (IPD) may be shared upon reasonable request. Access will be considered for qualified researchers with a valid scientific proposal. Requests will be reviewed by the study team, and a data sharing agreement may be required.

DOCUMENTS (1):
  • Study Protocol (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT07157475/Prot_000.pdf